CLINICAL TRIAL: NCT01959451
Title: Platelet Function Guided Prasugrel Therapy in ACS Patients Undergoing PCI
Brief Title: Testing Responsiveness to Platelet Inhibition on Chronic Antiplatelet Treatment For Acute Coronary Syndromes Trial
Acronym: TROPICAL-ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Dirk Sibbing, Prof. Dr. Dirk Sibbing, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MucT001-13
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Prasugrel; Clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel 5 mg or 10mg daily for 12 months.
  Interventions: Drug: Prasugrel
- Prasugrel/Clopidogrel (Experimental): Day 0 - 7 Prasugrel 5 or 10mg Day 8 - 14 Clopidogrel 75mg q/d. On Day 14 platelet function testing Patients with HPR will be switched to Prasugrel the others will remain on Clopidogrel for 11 1/2 months
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — see Arm description
  Other Names: Efient
  Arms: Prasugrel
Drug: Clopidogrel — see arm description
  Other Names: Iscover; Plavix
  Arms: Prasugrel/Clopidogrel

SUMMARY:
This study investigates whether a platelet function testing guided approach with a short-term (1 week) prasugrel treatment and a switch over to clopidogrel treatment in adequate responders to clopidogrel is non-inferior regarding the combined incidence of bleeding and thrombotic complications to a 12 month standard treatment with prasugrel in acute coronary syndrome (ACS) patients treated with percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Patients suffering of heart attack have highly activated blood platelets. During and after invasive treatment of blocked coronary vessels (percutaneous coronary intervention = PCI) a potent platelet inhibition is needed to reduce the risk of thrombotic complications which is particularly high within the first week after PCI. On the other hand, the use of potent platelet inhibitors such as prasugrel is associated with higher bleeding risk particularly when used at long-term. A combination of a potent antiplatelet drug (prasugrel) within the first week with a less potent antiplatelet drug (clopidogrel) thereafter might lead to a higher net clinical benefit - means less bleeding and thrombotic complications. This hypothesis is being investigated in the current trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Troponin positive ACS
* Successful PCI (defined as a post PCI diameter stenosis <20% and TIMI flow ≥2)
* A planned treatment of Prasugrel for 12 months after the procedure
* written informed consent

Exclusion Criteria:

* Age <18 years and >80 years
* Subjects with known contraindications to Clopidogrel treatment, which are hypersensitivity to the drug substance or any component of the product and active pathological bleeding such as peptic ulcer or intracranial hemorrhage
* Subjects with known contraindications to Prasugrel treatment, which are hypersensitivity to the drug substance or any component of the product, active pathological bleeding such as peptic ulcer or intracranial hemorrhage and a history of prior transient ischemic attack (TIA) or stroke
* Cardiogenic shock
* Subjects requiring concomitant treatment with an anticoagulant agent (Vitamin-K antagonists or novel oral anticoagulants such as Rivaroxaban, Dabigatran or Apixaban)
* Indication for major surgery (per decision of the treating physician) for the planned duration of the study
* Simultaneous participation in another clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to clinical trial beginning
* Known or persistent abuse of medication, drugs or alcohol
* Current or planned pregnancy or nursing women, women 90 days after childbirth. Females of childbearing potential, who do not use and are not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases
* Evidence of significant active neuropsychiatric disease, in the investigator's opinion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Composite of death from cardiovascular cause, myocardial infarction, stroke and bleeding grade ≥ 2 defined according to BARC criteria | 12 months

SECONDARY OUTCOMES:
bleeding events BARC class ≥2 | 12 months
stent thrombosis | 12 months
all-cause death | 12 months

OTHER OUTCOMES:
economic impact of a platelet function testing guided tailored treatment for ACS patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Sibbing, MD, Principal Investigator — Munich University Hospital; Julinda Mehilli, MD, Principal Investigator — Munich University Hospital; Steffen Massberg, MD, Study Chair — Munich University Hospital
Locations (33):
- Austria (2):
  - Medizin-Universität Graz, Univ. Klinik für Innere Medizin, Graz
  - Wilhelminenspital Wien, 3. Medizinische Abteilung, Vienna
- Germany (20):
  - Klinikum Augsburg, Department of Cardiology, Augsburg
  - Heart Center Bad Krozingen, Bad Krozingen
  - Asklepios Stadtklinik Bad Tölz, Internal Medicine, Bad Tölz
  - St. Josef Hospital, Katholisches Klinikum Bochum, Department of Cardiology, Bochum
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Frankfurt, Department of Cardiology, Frankfurt
  - Kliniken Ostallgäu-Kaufbeuren, Klinik Füssen, Füssen
  - Heart Center at the University Medical Center Goettingen, Göttingen
  - Universitätsmedizin Greifswald, Klinik u. Poliklinik für Innere Medizin B, Greifswald
  - Universitäres Herzzentrum Hamburg, UKE, Hamburg
  - University Hospital Mainz, Department of Cardiology, Mainz
  - Klinikum Memmingen, Innere Medizin I, Memmingen
  - Munich University Hospital, Munich
  - Klinikum Neuperlach, Department of Cardiology, Munich
  - Klinikum Bogenhausen, Department of Cardiology, Munich
  - Klinikum Oldenburg gGmbH, Herz-Kreislauf-Zentrum, Klinik für Kardiologie, Oldenburg
  - Universitätsmedizin Rostock, Zentrum für Innere Medizin, Rostock
  - Helios-Klinikum Siegburg, Abteilung für Kardiologie und Angiologie, Siegburg
  - University Hospital of Tuebingen, Department of Cardiology, Tübingen
  - Kliniken Nordoberpfalz AG, Klinikum Weiden, Medizinische Klinik II, Weiden
- Hungary (7):
  - Semmelweis Egyetem Kardiovaszkuláris Centrum, Budapest
  - Budapest Military Hospital, Budapest
  - Heart Center Balatonfüred, Budapest
  - Department of Cardiology Petz Aladár Megyei Oktató Kórház, Győr
  - Heart Center Kecskemet, Kecskemét
  - PTE KK Szívgyógyászati Klinika Intervenciós Kardiológia Részleg, Pécs
  - Heart Center Szeged, Szeged
- Poland (4):
  - 3rd Department of Cardiology, Upper Silesian Medical Centre, Medical University of Silesia, Katowice, Katowice
  - 1st Department of Cardiology, Poznan University of Medical Science, Poznan
  - 1st Department of Cardiology, Medical University of Warsaw, Warsaw
  - Department of Interventional Cardiology and Angiology, Institute of Cardiology, Warsaw, Warsaw

REFERENCES:
- [Derived] Sibbing D, Aradi D, Jacobshagen C, Gross L, Trenk D, Geisler T, Orban M, Hadamitzky M, Merkely B, Kiss RG, Komocsi A, Dezsi CA, Holdt L, Felix SB, Parma R, Klopotowski M, Schwinger RHG, Rieber J, Huber K, Neumann FJ, Koltowski L, Mehilli J, Huczek Z, Massberg S; TROPICAL-ACS Investigators. Guided de-escalation of antiplatelet treatment in patients with acute coronary syndrome undergoing percutaneous coronary intervention (TROPICAL-ACS): a randomised, open-label, multicentre trial. Lancet. 2017 Oct 14;390(10104):1747-1757. doi: 10.1016/S0140-6736(17)32155-4. Epub 2017 Aug 28. PMID 28855078
- [Derived] Sibbing D, Aradi D, Jacobshagen C, Gross L, Trenk D, Geisler T, Orban M, Gori T, Hadamitzky M, Merkely B, Kiss RG, Komocsi A, Dezsi CA, Thalmeier A, Low A, Holdt L, Teupser D, Ince H, Felix SB, Parma R, Malek L, Horstkotte J, Baylacher M, Schwinger R, Rieber J, Mudra H, Hausleiter J, Huber K, Neumann FJ, Koltowski L, Huczek Z, Mehilli J, Massberg S; TROPICAL-ACS Investigators. A randomised trial on platelet function-guided de-escalation of antiplatelet treatment in ACS patients undergoing PCI. Rationale and design of the Testing Responsiveness to Platelet Inhibition on Chronic Antiplatelet Treatment for Acute Coronary Syndromes (TROPICAL-ACS) Trial. Thromb Haemost. 2017 Jan 5;117(1):188-195. doi: 10.1160/TH16-07-0557. Epub 2016 Sep 22. PMID 27652610
- See also: Rationale and design of the Testing Responsiveness to Platelet Inhibition on Chronic Antiplatelet Treatment for Acute Coronary Syndromes (TROPICAL-ACS) Trial — http://www.ncbi.nlm.nih.gov/pubmed/27652610